CLINICAL TRIAL: NCT01670240
Title: Adalimumab (Humira) in the Treatment of Chronic Pouchitis
Brief Title: Adalimumab in the Treatment of Chronic Pouchitis
Acronym: ADAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Hvidovre University Hospital (Other); Aarhus University Hospital (Other); AbbVie (Industry)
Responsible Party: Principal Investigator, Mie Dilling Kjaer, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-004268-31
Record Dates: First submitted 2012-08-08; First posted 2012-08-22 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Ulcerative Colitis; Pouchitis
Keywords: IPAA; Pouchitis; Ulcerative colitis; Pouch; Adalimumab; Humira
MeSH Terms: conditions — Colitis, Ulcerative; Pouchitis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab (Active Comparator): Every second week, mg: 160-80-40-40-40-40 12 weeks in all
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Given as the active comparator, every second week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab
  Other Names: Humira
  Arms: Adalimumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study wants to investigate the efficiency of biological treatment for chronic pouchitis. Chronic pouchitis is inflammation in a reconstruction after removal of the colon, a pouch. It is examined in patients with ulcerative colitis.

The primary objective evaluation is to evaluate the clinically effect of biological therapy (adalimumab) in patients with chronic pouchitis.

Secondary objective is to evaluate the effect of biological therapy on the endoscopical and histological inflammatory activity.

It is a double-blinded randomized placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Operated with proctocolectomy and construction of an IPAA
* Prior to surgery diagnosed with ulcerative colitis according to established clinically, radiologic, endoscopic and histological criteria.
* Diagnosed with chronic pouchitis as defined above
* PDAI ≥ 7, with the clinically part of PDAI >2 and the endoscopic part of PDAI >3
* Age >18 years
* Negative stool cultures for bacterial bowel pathogens and negative stool microscopy for parasites
* Serology negative for chronic hepatitis B
* Negative examination for tuberculosis (including x-ray of thorax and a interferon gamma test)
* Signed informed consent

Exclusion Criteria:

* Treatment with glucocorticoids within the last 4 weeks
* Diagnosed with Crohn's disease
* Need of an interpreter or if patients do not understand oral or written information.
* Surgical complications as anal stenosis, leak of the anastomosis, or fistula arising from the pouch
* Abuse of medicine, alcohol or drugs
* Ongoing treatment with NSAID (non steroid anti inflammatory drug)
* Pregnancy or nursing
* A diverting stoma
* Malignancy or other severe chronic disease or expected longevity less than one year
* Patients diagnosed with immune deficiency
* Ongoing infectious disease
* Contraindications against treatment with tumor necrosis factor-alpha antibody, such as heart disease, former cancer disease, in vivo vaccination within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinical response on treatment with Adalimumab | 12 weeks
  The number of patients with chronic pouchitis achieving a clinical improvement, defined as a reduction in clinically PDAI ≥ 2 at any time within the 12 weeks of treatment with adalimumab (Humira).
  Clinical PDAI (0-6 points)(pouchitis disease activity index)refers to fewer (0-1 point), number of bowel movements(0-2 points), rectal bleeding(0-1 point) and fecal urgency(0-2 points).

SECONDARY OUTCOMES:
Clinical improvement after 12 weeks of treatment | 12 weeks
  The number of patients with a clinical improvement (PDAI reduction ≥ 2)at week 12 See the description of clinical improvement and PDAI under primary endpoint
Clinical remission after 12 weeks | 12 weeks
  The number of patients with pouchitis in remission at week 12 (total PDAI ≤4)
Endoscopic and histologic response after treatment with Adalimumab | 12 weeks
  Effect (reduction in PDAI)of adalimumab (Humira) on the endoscopical and histological activity in chronic pouchitis Endoscopical and histological activity is defined from PDAI (pouchitis disease activity index). Endoscopically the presence of Edema, Granularity, Friability, Loss of vascular pattern, Mucous exudates or Ulceration, gives 1 point each (max 6 points). Histological the presence of polymorphic nuclear leukocyte infiltration and ulceration each gives 1-3 points regarding severity (max 6 points)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kjeldsen, Phd, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark